CLINICAL TRIAL: NCT01838265
Title: A Randomized Two-Arm Trial of Prostate Cancer Patients Undergoing Active Surveillance With or Without MRI-Guided Management: The MGM Trial
Brief Title: Trial of Prostate Cancer Patients Undergoing Active Surveillance With or Without MRI-Guided Management
Acronym: MGM
Status: Withdrawn | Type: Observational
Why Stopped: Unlikely to Accrue
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Sanoj Punnen, Assistant Professor, University of Miami
Other Study IDs: 20120698
Record Dates: First submitted 2013-04-18; First posted 2013-04-24 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Biomarkers; Hematologic Tests; Blood Urea Nitrogen; Creatinine; Prostate-Specific Antigen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsy tumor tissue, blood and urine samples for correlative studies (circulating tumor cells (CTC), free-circulating DNA (fcDNA) and single nucleotide polymorphisms (SNPs)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- AS: Active Surveillance Alone: Active Surveillance Alone (AS). Transrectal Ultrasound-guided biopsies within 6 months of enrollment and at 1 year intervals thereafter (maximum four biopsies).
  Interventions: Procedure: Transrectal Ultrasound-Guided Biopsy; Behavioral: Expanded Prostate Cancer index Composite Questionnaire; Behavioral: Short-Form 12 of Health Related Quality of Life Questionnaire; Behavioral: Memorial Anxiety Scale for Prostate Cancer; Procedure: Plasma/Serum Sample for biomarkers; Procedure: Urine Sample for Biomarkers; Procedure: Blood Tests for Blood Urea Nitrogen and Creatinine; Procedure: Blood Test for Serum PSA
- MRI-AS: MRI+ Active Surveillance: MRI-Managed Active Surveillance (MRI-AS). MRI Ultrasound or MRI-guided biopsies within 6 months of enrollment and at 1 year intervals thereafter (maximum four biopsies)
  Interventions: Procedure: MRI Ultrasound Biopsy; Behavioral: Expanded Prostate Cancer index Composite Questionnaire; Behavioral: Short-Form 12 of Health Related Quality of Life Questionnaire; Behavioral: Memorial Anxiety Scale for Prostate Cancer; Procedure: Plasma/Serum Sample for biomarkers; Procedure: Urine Sample for Biomarkers; Procedure: Blood Tests for Blood Urea Nitrogen and Creatinine; Procedure: Blood Test for Serum PSA

INTERVENTIONS:
Procedure: Transrectal Ultrasound-Guided Biopsy — Active Surveillance Alone (AS). Transrectal Ultrasound-guided biopsies within 6 months of enrollment and at 1 year intervals thereafter (maximum four biopsies).
  Other Names: TRUS
  Groups: AS: Active Surveillance Alone
Procedure: MRI Ultrasound Biopsy — MRI-Managed Active Surveillance (MRI-AS). MRI Ultrasound or MRI-guided biopsies within 6 months of enrollment and at 1 year intervals thereafter (maximum four biopsies)
  Groups: MRI-AS: MRI+ Active Surveillance
Behavioral: Expanded Prostate Cancer index Composite Questionnaire — Quality of life questionnaire obtained at Baseline, and at 12, 24 and 36 months after initial biopsy
  Other Names: EPIC
Behavioral: Short-Form 12 of Health Related Quality of Life Questionnaire — Quality of life questionnaire obtained at Baseline, and at 12, 24 and 36 months after initial biopsy
  Other Names: SF-12; SF-12 HRQOL
Behavioral: Memorial Anxiety Scale for Prostate Cancer — Quality of life questionnaire obtained at Baseline, and at 12, 24 and 36 months after initial biopsy
  Other Names: MAX-PC
Procedure: Plasma/Serum Sample for biomarkers — Plasma/Serum Sample for biomarkers obtained at Baseline, and at 12, 24 and 36 months after initial biopsy for correlative studies (CTC, fcDNA, SNPs)
Procedure: Urine Sample for Biomarkers — Urine Sample for biomarkers obtained at Baseline, and at 12, 24, and 36 months for correlative studies (hypermethylated DNA)
Procedure: Blood Tests for Blood Urea Nitrogen and Creatinine — Blood Tests for Blood Urea Nitrogen (BUN) and Creatinine obtained at 0 - 6 months, and at 12, 24, and 36 months from initial biopsy. This is optional, subject may refuse
Procedure: Blood Test for Serum PSA — Blood test for Serum PSA obtained at Baseline, at every 6 months up to 36 months from initial biopsy.
  Other Names: PSA test

SUMMARY:
1. Using multiparametric MRI Ultrasound-guided or MRI-guided biopsies will allow more accurate sampling of the tumors and therefore will increase the rate of "progression" on early (first and second) surveillance biopsies and decrease the rate of "progression" on late (third and further) surveillance biopsies compared to Transrectal Ultrasound-guided biopsies.
2. Quality of life (QoL) will be similar in patients undergoing MRI Ultrasound or MRI-guided and Transrectal Ultrasound-guided biopsies.
3. Biomarker expression levels will correlate with biopsy progression.

DETAILED DESCRIPTION:
Favorable risk patients will be randomized to one of two active surveillance arms. Stratification will be based on Prostate-specific antigen density (PSAD) (=< 0.15 vs > 0.15 ng/mL per mL), and number of positive cores in the diagnostic biopsy (1 vs 2):

* Arm I: Active Surveillance Alone (AS). TRUS guided biopsies at start (within 6 months of enrollment) and at yearly intervals thereafter up to 36 months after the initial biopsy (maximum four biopsies).
* Arm II: MRI-Managed Active Surveillance (MRI-AS). MRIus or MRI-guided biopsies at start (within 6 months of enrollment) and at yearly intervals thereafter up to 36 months after the initial biopsy (maximum four biopsies).

Patients will also complete Quality of Life (QoL) assessments to provide unique data on the effects of MRI monitoring for patients undergoing active surveillance on QOL. The investigators have selected a group of measures that have been used extensively in prostate cancer populations.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed adenocarcinoma of the prostate.
* Biopsy must consist of at least 8 cores.
* Enrollment is =< 1 year from diagnosis.
* One or two biopsy cores with less than 50% tumor present in each core and Gleason score =< 6 (3+3).
* Candidate for multiparametric MRI.
* T1-T2a disease based on digital rectal exam.
* No concurrent, active malignancy, other than nonmetastatic skin cancer or early stage chronic lymphocytic leukemia (well-differentiated small cell lymphocytic lymphoma). If a prior malignancy is in remission for >= 5 years then the patient is eligible.
* Ability to understand and willingness to sign a written informed consent document
* Zubrod performance status < 2.
* Patients must agree to fill out the psychosocial questionnaires.
* Age >= 35 and =< 75 years

Exclusion Criteria:

* Not biopsy confirmed adenocarcinoma of the prostate.
* Biopsy consists of less than 8 cores.
* Three or more biopsy cores are positive.
* Gleason score >= 3+4=7.
* A single core has >= 50% involvement with Gleason score =6 (3+3) or less.
* DCE-MRI study before enrollment.
* Inability to undergo MRI exam.
* Greater than T2a disease based on digital rectal exam.
* Concurrent, active malignancy, other than nonmetastatic skin cancer or early stage chronic lymphocytic leukemia (well-differentiated small cell lymphocytic lymphoma). If a prior malignancy is in remission for < 5 years then the patient is ineligible
* Inability to understand or unwilling to sign a written informed consent document.
* Zubrod performance status >= 2.
* Patient unwilling to fill out the psychosocial questionnaires.
* Age < 35 or > 75.

Ages: 35 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Low risk male patients with early stage T1 - T2a prostate adenocarcinoma, based on a digital rectal exam palpation. Patients must also have less than three positive cores with < 50% of a single core; and Gleason score 3 + 3 = 6 or less.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Rate of Progression in Subjects undergoing MRIus Biopsy vs Standard Ultrasound biopsy | 42 months
  To determine of multiparametric MRIus-guided biopsies increase the rate of progression on early (first two) biopsies in men undergoing active surveillance as compared with early detection using standard ultrasound biopsy.

SECONDARY OUTCOMES:
Expression Levels of Biomarkers from biopsies collected with MRI-us Biopsy vs Standard Ultrasound Biopsy | 42 months
Effect of MRI Monitoring on Health-Related Quality of Life | 42 months
  To determine the effect of MRI monitoring on health-related quality of life (HRQOL), prostate cancer-specific anxiety QOL (ie general, PSA-testing & recurrence anxiety, PC-Anxiety) and prostate cancer-specific QOL (ie sexual, urinary & bowel function, PC-QOL), particularly as they relate to ethnically and socioeconomically diverse and disparate populations.

CONTACTS AND LOCATIONS:
Overall Officials: Dipen Parekh, MD, Principal Investigator — University of Miami; Alan Pollack, MD, Principal Investigator — University of Miami; Sanoj Punnen, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States